CLINICAL TRIAL: NCT02334332
Title: Pilot Study of an Educational Brochure to Prepare Patients and Informal Caregivers for Recovery Following Gastrectomy
Brief Title: Educational Brochure in Preparing Patients With Gastric Cancer and Their Caregivers for Recovery After Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No accrual
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14286; NCI-2014-02563 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14286 (Other: City of Hope Medical Center)
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Anxiety; Gastric Carcinoma; Stress
Keywords: Caregiver
MeSH Terms: conditions — Anxiety Disorders; Stomach Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort I (standard care) (Active Comparator): Participants receive standard post-operative care.
  Interventions: Procedure: Standard Follow-Up Care; Procedure: Quality-of-Life Assessment
- Cohort II (educational brochure) (Experimental): Participants receive a 2-page educational brochure after surgery and prior to discharge home.
  Interventions: Other: Educational Intervention; Procedure: Quality-of-Life Assessment

INTERVENTIONS:
Other: Educational Intervention — Receive educational brochure
  Other Names: Education for Intervention; Intervention, Educational
  Arms: Cohort II (educational brochure)
Procedure: Standard Follow-Up Care — Receive standard post-operative care
  Arms: Cohort I (standard care)
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot clinical trial studies an educational brochure in preparing patients with gastric cancer and their caregivers for recovery after surgery. Giving an educational brochure may help prepare patients and their caregivers by improving knowledge about symptoms after surgery. It may also improve quality of life and reduce worry after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To pilot test an educational intervention in the form of a teaching brochure to prepare patients and informal caregivers for recovery following partial or total gastrectomy.

SECONDARY OBJECTIVES:

I. To describe preliminary effect of the intervention on patient-reported outcomes (PROs), informal caregiver-reported outcomes, and clinical/system outcomes.

OUTLINE: Participants are enrolled sequentially to 1 of 2 cohorts.

COHORT I: Participants receive standard post-operative care.

COHORT II: Participants receive a 2-page educational brochure after surgery and prior to discharge home.

After completion of study, participants are followed up for approximately 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be accrued using the following inclusion criteria:

  * Scheduled to undergo partial or total gastrectomy for treatment of gastric cancer
  * Able to read and understand English
* Informal Caregivers will be accrued using the following inclusion criteria:

  * The primary informal caregiver as identified by patients participating in the study; this refers to either a family member or friend who will be providing the majority of care following surgery
  * Able to read and understand English
* All participants must have the ability to understand the willingness to provide informed consent

Exclusion Criteria:

* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Patient/informal caregiver satisfaction with timing, content, and delivery of the intervention | Up to 2 months
  Descriptive statistics will be presented through summary statistics of data from the satisfaction tools.

SECONDARY OUTCOMES:
Change in mean survey scores | Baseline up to 4 weeks
  Data will be summarized using descriptive statistics. Statistics will be tabulated for each sequentially enrolled cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States